CLINICAL TRIAL: NCT03607409
Title: Role of Inhibin A as Biomarker for Ovarian Response to Stimulation With Gonadotropins for IVF Treatment
Brief Title: Role of Inhibin A as Biomarker for Ovarian Response for IVF Treatment
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: Ansh Labs (Unknown)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 1806-ABU-043-BL
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the role of Inhibin A as bio marker for the number of mature oocytes, compared to Estradiol

DETAILED DESCRIPTION:
Inhibin A could be an improved biomarker regarding the number of expected mature oocytes compared to estradiol.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing ovarian stimulation with gonadotropins in either a GnRH-agonist or GnRH-antagonist for IVF treatment due to primary / secondary infertility.

Exclusion Criteria:

Patients undergoing a modified natural cycle stimulation protocol (Taymour cycle) Patients at risk for development of ovarian hyperstimulation syndrome (OHSS)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing ovarian stimulation for IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes | 1 year
  Patients undergoing ovarian stimulation with gonadotropins

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneyer AL, Fujiwara T, Fox J, Welt CK, Adams J, Messerlian GM, Taylor AE. Dynamic changes in the intrafollicular inhibin/activin/follistatin axis during human follicular development: relationship to circulating hormone concentrations. J Clin Endocrinol Metab. 2000 Sep;85(9):3319-30. doi: 10.1210/jcem.85.9.6767. PMID 10999828
- [Background] Hohmann FP, Laven JS, de Jong FH, Fauser BC. Relationship between inhibin A and B, estradiol and follicle growth dynamics during ovarian stimulation in normo-ovulatory women. Eur J Endocrinol. 2005 Mar;152(3):395-401. doi: 10.1530/eje.1.01871. PMID 15757856
- [Background] Abbara A, Vuong LN, Ho VNA, Clarke SA, Jeffers L, Comninos AN, Salim R, Ho TM, Kelsey TW, Trew GH, Humaidan P, Dhillo WS. Follicle Size on Day of Trigger Most Likely to Yield a Mature Oocyte. Front Endocrinol (Lausanne). 2018 Apr 25;9:193. doi: 10.3389/fendo.2018.00193. eCollection 2018. PMID 29743877